CLINICAL TRIAL: NCT00401167
Title: Phase IV-An Open-Label Prospective Study of Memantine in Institutionalized Patients With Severe Alzheimer's Disease and Significant Behavioural and Psychological Symptoms of Dementia
Brief Title: Memantine for Agitation and Aggression in Severe Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Lundbeck Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lundbeck-11267
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2010-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; behavioral and psychological symptoms of dementia; severe Alzheimer's disease; memantine; agitation; aggression
MeSH Terms: conditions — Alzheimer Disease; Behavior; Psychomotor Agitation; Aggression | interventions — Memantine

INTERVENTIONS:
Drug: memantine — Following the baseline visit, subjects will receive memantine 5 mg OD for one week, followed by 5 mg BID for one week, followed by 10 mg QAM and 5 mg QPM for one week, followed by 10 mg BID for the following 9 weeks.

SUMMARY:
Alzheimer's disease (AD) is the most common form of dementia and is characterized by both cognitive and behavioural symptoms ("Behavioural and Psychological Symptoms of Dementia"; BPSD). To date, there are only modestly effective treatments for BPSD, and these treatments are associated with an increased risk of mortality in elderly dementia patients. We plan to study whether treatment with medication memantine improves BPSD in severe AD patients. Thirty-two AD patients with significant BPSD, including agitation and aggression, will be treated for three months with memantine. Assessments of behavioural symptoms and global clinical outcomes will be completed after one, two and three months of treatment.

DETAILED DESCRIPTION:
BPSD in institutionalized patients with severe AD is a serious public health problem. The effectiveness of current pharmacological management of BPSD with atypical antipsychotics is modest at best, and there are serious safety concerns including increased cerebrovascular adverse events and increased mortality. Preliminary data with memantine suggests this medication may be helpful for treating BPSD in the severe subgroup of the Alzheimer's disease patient population. It is for this reason we propose an open-label prospective study of memantine in institutionalized patients with severe Alzheimer's disease and significant BPSD.

The major objective of this study is to examine the effectiveness of memantine on behaviour with a focus on agitation and aggression. The secondary objective is to determine the effect of memantine on nursing burden and prescription medication use. The study would expand clinical experience with memantine and provide information on professional caregiver burden and prescription medication use in this institutionalized, more severely impaired and frailer population. This information could be used to design a randomized placebo controlled confirmatory trial.

The effectiveness of memantine on agitation and aggression in patients with moderate to severe Alzheimer's disease will be assessed in a 3-month, open-label study involved 32 patients residing in long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from a legally acceptable representative
* Male or female > 65 years of age, residing in long-term care
* Diagnosis and Statistical Manual of Mental Disorders (DSM-IV-TR) diagnosis of Dementia of the Alzheimer's type (code 290.1)
* Mini Mental State Examination total score ≤ 15
* Neuropsychiatric Inventory-Nursing Home Version total score > 10, and a score > 1 on the agitation/aggression subscale
* A current order for any prescription medication for behavioral and psychological symptoms of dementia (e.g. benzodiazepine, antipsychotic, trazodone), with at least 1 dose used in the prior 3 months
* Patients with a current order for any regularly administered psychotropic (example, selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, trazodone, atypical antipsychotics, typical antipsychotics or cholinesterase inhibitors) must have been on a stable dose for 3 months prior to entry

Exclusion Criteria:

* Current evidence of any uncontrolled medical illness that would interfere with the subject's participation in the study
* Dementia due to any etiology other than Alzheimer's Disease
* Subjects experiencing significant difficulties ingesting oral medications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory Nursing Home Version | Screening, Baseline, 1 month, 2 months, 3 months
Clinical Global Impression of Change | Baseline, 1 month, 2 months, 3 months

SECONDARY OUTCOMES:
Neuropsychiatric Inventory Nursing Home Version | Screening, baseline, 1 month, 2 months, 3 months
Neuropsychiatric Inventory Burden Subscale | Screening, baseline, 1 month, 2 months, 3 months
Cohen Mansfield Agitation Inventory | Baseline, 1 month, 2 months, 3 months
Modified Nursing Care Assessment Scale | Baseline, 3 months
Activities of Daily Living | Baseline, 3 months
Quality of Life in Late Stage Dementia | Baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Herrmann, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - North York General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Result] Herrmann N, Cappell J, Eryavec GM, Lanctot KL. Changes in nursing burden following memantine for agitation and aggression in long-term care residents with moderate to severe Alzheimer's disease: an open-label pilot study. CNS Drugs. 2011 May;25(5):425-33. doi: 10.2165/11588160-000000000-00000. PMID 21476613